CLINICAL TRIAL: NCT03228030
Title: Thiamine Supplementation in Heart Failure: a Pilot Randomized Controlled Crossover Trial
Acronym: THIAMINE-HF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster/St. Peter's Hospital Chair of Aging (Unknown)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-387
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Thiamine Deficiency; Congestive Heart Failure
Keywords: thiamine; heart failure; heart failure with reduced ejection fraction; geriatric; thiamin; vitamin b1; congestive heart failure
MeSH Terms: conditions — Heart Failure; Thiamine Deficiency | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thiamine mononitrate 500mg po daily (Experimental): 3 months on thiamine, followed by 6 week washout period, and then 3 months on placebo arm
  Interventions: Dietary Supplement: Thiamine
- Placebo (Placebo Comparator): 3 months on placebo, followed by 6 week washout period, and then 3 months on thiamine
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Thiamine — Capsules
  Arms: Thiamine mononitrate 500mg po daily
Dietary Supplement: Placebo — Identical capsules
  Arms: Placebo

SUMMARY:
Heart failure (HF) is a major cardiovascular disease with increasing prevalence. Thiamine deficiency is common in HF patients. Previous small studies have shown that thiamine supplementation can improve left ventricular systolic function in HF, but larger clinical studies are lacking. Given the ease of supplementation and the potential benefits in HF, we aim to conduct a pilot randomized controlled trial (RCT) using high dose thiamine supplementation in HF patients. The main goal of this pilot study is to determine the feasibility of recruitment for an RCT of thiamine supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60
* NYHA class II-IV symptoms
* Recent HF-related admission in past 12 months OR NT-proBNP >600ng/L within 60 days of screening
* LVEF ≤45% on 2D/3D echocardiography or radionuclide angiography (RNA) in the past 12 months (on optimal therapy)
* Medically optimized prior to enrolment with angiotensin converting enzyme inhibitor or angiotensin receptor blocker (± neprilysin inhibitor), β-blocker, and/or aldosterone antagonist at target or maximally tolerated doses.
* Patients must be stable on medications without hospitalization in the past month.

Exclusion Criteria:

* Taking >2.5mg/d of thiamine supplement. Allows standard multivitamin. B complex vitamin not allowed due to high thiamine content.
* Unable to swallow study medication. A placebo swallowing test will take place at screening.
* Clinical indication for thiamine supplementation including symptomatic thiamine deficiency (Wernicke's encephalopathy, severe malnutrition, refeeding syndrome) and heavy alcohol use, >15 standard drinks per week in men and >10 standard drinks per week in women.
* End-stage renal disease on dialysis
* Severe mitral valve disease because this impacts the accuracy of speckle tracking analysis on echocardiography.
* Non-English speaking (unable to complete questionnaires).
* Unable to provide written consent.
* Cognitive impairment without a caregiver administering medications.
* Expected survival <1 year due to non-cardiac disease.
* Expected heart transplantation in <6 months (± left ventricular assistive device).
* Allergies to the ingredients of the study medication or placebo

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Recruitment | 11 months
  Number of participants recruited during the study period. This is a feasibility outcome.

SECONDARY OUTCOMES:
Refusal rate | 11 months
  Number of eligible individuals refusing to participate in the research study. This is a feasibility outcome
Retention rate | 11 months
  Number of participants completing the study.
Compliance rate | 11 months
  Proportion of participants with >80% adherence to intervention.
Left ventricular ejection fraction (LVEF) | 3 months
  Echocardiogram measurement of left ventricular ejection fraction.
Peak global longitudinal strain (%) | 3 months
  Speckle tracking echocardiogram measurement of heart contractility. This is a more sensitive measurement of heart function than LVEF.
NT-proBNP | 3 months
  Heart failure biomarker
New York Heart Association (NYHA) class | 3 months
  Heart function symptom grading
Quality of life | 3 months
  Kansas City Cardiomyopathy Questionnaire
HF hospitalizations | 7.5 months
  Number of hospital stays >24h
HF emergency room visits | 7.5 months
  Number of hospital visits <24h
Death due to cardiovascular causes | 7.5 months
  As adjudicated by study committee

CONTACTS AND LOCATIONS:
Overall Officials: Eric KC Wong, MD FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wong EKC, Lee JY, Leong DP, Mbuagbaw L, Yousuf H, Keen S, Straus SE, Patterson CJ, Demers C. Thiamine versus placebo in older heart failure patients: study protocol for a randomized controlled crossover feasibility trial (THIAMINE-HF). Pilot Feasibility Stud. 2018 Sep 20;4:149. doi: 10.1186/s40814-018-0342-0. eCollection 2018. PMID 30258648